CLINICAL TRIAL: NCT06222021
Title: Hyperlactacidemia in Major Abdominal Surgery: Role of Variation in the Monocarboxylate Receptors
Brief Title: Hyperlactacidemia in Major Abdominal Surgery and Monocarboxylate Receptors
Acronym: NETTUNO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 5675
Record Dates: First submitted 2024-01-02; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2023-12

CONDITIONS: Surgical Procedure, Unspecified; Postoperative Complications; Hyperlactatemia; Abdomen Disease
MeSH Terms: conditions — Postoperative Complications; Hyperlactatemia

STUDY DESIGN:
Intervention Model Description: Participants will undergo preoperative genomic assay testing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Genetic analysis of polymorphisms of membrane receptors involved in lactate transport (Other): Before the start of surgery, after arterial line cannulation, a blood sample will be collected in an ethylenediaminetetraacetic acid (EDTA) test tube for genetic analysis of polymorphisms of membrane receptors involved in lactate transport including transporter family monocarboxylates 1 (MTC1), transporter family monocarboxylates 4 (MTC4) and Gi-coupled protein receptor 81 (GPR81).
  Interventions: Genetic: Genetic analysis of polymorphism of membrane receptors involved in lactate transport

INTERVENTIONS:
Genetic: Genetic analysis of polymorphism of membrane receptors involved in lactate transport — The DNA extracted from the blood samples (through extractor MagCore) will then undergo gene sequencing by Sanger sequencing and/or Custom NGS (Next Generation Sequencing) panels and will be used to identify nucleotide variants within genes involved in lactate transport (MCT-1/4, GPR81).

SUMMARY:
The goal of this clinical trial is to identify those situations in which the increase of lactate levels is not clinically relevant since it is associated with altered genetic polymorphism of the genes involved in the membrane proteins acting as carriers for lactate (mainly monocarboxylate transporters, MCTs) patients undergoing major abdominal surgery.

The main questions it aims to answer are:

1. Is there a relationship between the lactate levels in the immediate post-operative period and the presence of some lactate receptor polymorphisms?
2. Can hyperlactacidemia related to lactate receptor polymorphisms affect length of stay in the recovery room and/or in intensive care unit, postoperative hospital stay, postoperative complications? - Which are the risk factors for hyperlactacidemia in the immediate post-operative period in addition to the presence of lactate receptors polymorphisms?

Participants will undergo pre-operative genomic assay testing.

DETAILED DESCRIPTION:
Lactic acidosis is traditionally attributed to cellular hypoxia, to an imbalance between the body's demand for oxygen and its availability. Lactate is produced by the muscles, skin, brain, red blood cells and intestine and eliminated by the liver and kidneys. Lactate is produced by the following biochemical reaction: Pyruvate + reduced nicotinamide adenine dinucleotide (NADH) + H+ ↔ Lactate + nicotinamide-adenine dinucleotide (NAD+). Under normal conditions, this reaction produces lactate from pyruvate in a ratio of 10 to 1. Pyruvate comes from glycolysis and is used by mitochondria. When glycolysis is increased or mitochondrial oxidative phosphorylation is blocked, pyruvate accumulates and is converted into lactate generating hyperlactacidemia and acidosis. Normal lactate levels are 0-2 mmol/L. Hyperlactacidemia, usually defined as values above 2.2 mmol/L, is divided into two types: A (associated with hypoxia) and B (related to increased stress-induced aerobic metabolism, mitochondrial diseases and the use of drugs such as metformin and beta2 agonists). The lactate/pyruvate ratio allows us to distinguish the two types of hyperlactacidemia. In hyperlactacidemia type A, this ratio is >10 while in type B it remains constant (L/P=10). In case of liver dysfunction, hyperlactacidemia may be associated with a variable L/P ratio based on the determining cause reduction in lactate clearance. In fact, lactate extraction may depend on the hepatic blood flow, the polymorphism of some genes involved in the lactate transport (mainly MCT1) and the potential of hydrogen (pH) which inhibits gluconeogenesis when lower than 7.10. Since lactic acid is an hydrophilic weak acid, its transport across membranes requires transporters that belong to the transporter family monocarboxylates (MCTs) encoded by the solute carrier family 16 (SLC16) gene family. It has been demonstrated that the MCT1 (rs1049434) T1470A polymorphism is associated with a deficit in the transmembrane transport of lactate: in fact, the T allele is correlated with an approximately 50% reduction in the lactate transport rate compared to the A6 allele. MCT4, which has a very low affinity for pyruvate and a greater affinity for lactate, ensures that pyruvate is converted into lactate before transmembrane transport. Polymorphisms affecting these receptors can influence the different speed of transmembrane lactate flow and therefore correlate with lesser or greater accumulation of serum lactate. Another membrane receptor involved in lactate transport has recently been described: G-coupled protein receptor 81 (GPR81), present in adipocytes. Polymorphisms affecting the gene encoding this receptor could correlate with a different accumulation of lactate. An increase in the level of lactates is often correlated with increased morbidity and mortality in critical situations critical such as sepsis, trauma, major cardiac and abdominal surgery. Measurement of perioperative biomarkers such as lactate is often used in clinical practice as an outcome predictor. However, there are no studies aimed to identify those situations in which the increase of lactates is not clinically relevant since it is associated with altered genetic polymorphism.

The investigators hypothesized that lactate levels at 3 hours after the end of major abdominal surgery will be higher in the patients carrying the T allele versus the A allele for MCT1 gene.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Indication for elective major abdominal surgery

Exclusion Criteria:

* Age <18 years
* Liver cirrhosis
* Liver surgery
* Intraoperative chemotherapy
* Previous gastric bypass surgery (thiamine deficiency)
* Severe cardiovascular/respiratory impairment
* Mitochondrial diseases
* Pheochromocytoma
* Chronic renal failure ≥ stage III
* Refusal to sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Lactate levels | 3 hours after the end of surgery
  Lactate levels (mmol/L) in the patients carrying the T allele versus the A allele for MCT1 gene.

SECONDARY OUTCOMES:
Polymorphisms of lactate receptors (presence of MCT4 and GPR8) | Minutes and an average of 30 minutes before the start of surgery
  Prevalence of the lactate receptors MCT4 and GPR8 polymorphisms throughout the genetic analysis of a blood sample.
Lactate clearance | 3 hours after the end of surgery
  Evaluation of the association between lactate clearance (lactate levels at the end of surgery - lactate levels at 3 hours after the end of surgery)x100/lactate levels at the end of surgery and the presence of lactate receptor polymorphisms (MCT4 and GPR8).
Lactate clearance | 24 hours after the end of surgery
  Evaluation of the association between lactate clearance (lactate levels at the end of surgery - lactate levels at 24 hours after the end of surgery)x100/lactate levels at the end of surgery and the presence of lactate receptor polymorphisms (MCT4 and GPR8).
Postoperative recovery | Hours (RR) or days (ICU) and average of three hours for RR and one day in ICU
  Length of stay in recovery room (RR) or in intensive care (ICU)
In-hospital stay | Days until discharge, an average of 7 day
  Hospital stay duration
Hyperlactacidemia | 3 hours after the end of surgery
  Analysis of potential risk factors for hyperlactacidemia (lactate levels >2.2 mmol/L) as well as the presence of lactate receptor polymorphisms including age (years), comorbidities, American Society of Anesthesiologists (ASA) physical status classification system, Body Mass Index (kg/m2), type and duration of surgery (hours), surgical approach (open, laparoscopic, robotic), total of liquids administered (ml), total diuresis (ml), blood losses (ml), intraoperative blood components transfusions (units), blood gas analyses parameters, number of hypotensive episodes during surgery (MAP<65 mmHg) requiring the administration of norepinephrine or its dosage increase.

CONTACTS AND LOCATIONS:
Locations (1):
- UOC Anestesia delle Chirurgie Generali e dei Trapianti, Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Italy/Lazio, Italy